CLINICAL TRIAL: NCT03546270
Title: The Effects of Swimming Training on Arterial Function, Strength and Cardiorespiratory Capacity in Elderly Women With Stage 2 Hypertension
Brief Title: The Effects of Swimming on Elderly Women With Stage-2 Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University (Other)
Collaborators: Marymount University (Other); Dong-Eui University (Other); University of Nebraska (Other)
Responsible Party: Principal Investigator, Won-mok son, Principal Investigator, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SwimmingMenopause
Record Dates: First submitted 2018-05-22; First posted 2018-06-06 (Actual); Results first posted 2019-08-05 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Menopause; Hypertension
Keywords: Swimming; Arterial Stiffness; Blood Pressure; Muscular Strength; Cardiorespiratory Endurance
MeSH Terms: conditions — Hypertension | interventions — Swimming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swimming (Experimental): Participants performed SWM training (combination of free style, breast stroke, and backstroke) for 20 weeks. For the first 5 weeks subjects swam 25-30 minutes/day, 3-4 days/week at ~60% of maximal heart rate. As their overall level of fitness and exercise skill improved, the intensity and duration of exercise increased to 40-45 minutes/day, 3-4 days/week at an intensity of 70-75% of the HRmax. Target HR was adjusted based on the observation that maximal heart rate during SWM is approximately 12 beats/min lower than that during running. Each subject was instructed to swim continuously except during the time needed for checking a target heart rate
  Interventions: Behavioral: Swimming
- Control (No Intervention): Participants in the non-exercising control group did not participate in a supervised exercise program and visited the laboratory at the same frequency as participants in the swim intervention and underwent recreational activities such as board games

INTERVENTIONS:
Behavioral: Swimming — This group completed 20-weeks of swimming
  Arms: Swimming

SUMMARY:
Aging is associated with progressive decreases in arterial health and function as well as overall fitness. It is crucial to prevent or reduce the negative effects of aging on the vasculature and fitness components by implementing appropriate lifestyle interventions, such as exercise training. We examined the effects of a swimming (SWM) regimen on arterial stiffness (pulse wave velocity, PWV), blood pressure (BP), wave reflection (AIx), muscle strength and aerobic capacity in elderly women with stage 2 hypertension.

DETAILED DESCRIPTION:
Using a parallel experimental design, participants were randomly assigned to either SWM (n=52) or non-exercising control group (n=48) for 20 weeks. Participant in the SWM group trained 3-4 days/week, progressing in duration from 25 to 45 min. Participants' carotid to radial PWV (crPWV), systolic and diastolic BP, AIx, strength and VO2max were measured at baseline and after 20 weeks of their assigned intervention.

ELIGIBILITY:
Inclusion Criteria:

* systolic/diastolic BP: 140-179 over 90-119 mm Hg
* had experienced the absence of menstruation for at least 1 year
* body mass index <30 kg/m2
* <1 h of regular exercise per week in the previous year

Exclusion Criteria:

* Smoker
* Taking any medications or hormone therapy in previous year

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-04 (Actual)

REFERENCES:
- [Derived] Wong A, Kwak YS, Scott SD, Pekas EJ, Son WM, Kim JS, Park SY. The effects of swimming training on arterial function, muscular strength, and cardiorespiratory capacity in postmenopausal women with stage 2 hypertension. Menopause. 2018 Dec 17;26(6):653-658. doi: 10.1097/GME.0000000000001288. PMID 30562322

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Swimming | Control
Started | 52 | 48
Completed | 52 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Swimming | Control | Total
Number analyzed (Participants) | 52 | 48 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (4) | 73 (4) | 74 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 48 | 100
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 52 | 48 | 100
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Pressure wave reflection [Mean (Standard Deviation); unit: percent] — augmentation index (percentage of pressure wave reflection), normalized to 75bpm
  percent | 31 (3) | 30 (2) | 31 (3)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 146 (1.7) | 144 (1) | 145 (1.4)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 88 (1.7) | 91 (1) | 90 (1.4)
Arterial stiffness [Mean (Standard Deviation); unit: m/s] — carotid-to-radial pulse wave velocity
  m/s | 9.0 (0.2) | 9.4 (0.2) | 9.2 (0.2)
Muscular strength [Mean (Standard Deviation); unit: kg] — hand grip dynamometry
  kg | 24 (1) | 25 (1) | 25 (1)
Cardiorespiratory endurance [Mean (Standard Deviation); unit: mL/kg/min] — Bruce treadmill test, VO2max
  mL/kg/min | 22 (2) | 24 (3) | 23 (3)

OUTCOME MEASURES:

1. Primary Outcome: Arterial Stiffness
Description: via Pulse Wave Velocity
Time Frame: 20-weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Swimming | Control
Number analyzed (Participants) | 52 | 48
m/s | 7.8 (0.3) | 10.0 (0.2)

2. Secondary Outcome: Systolic Blood Pressure
Description: systolic blood pressure
Time Frame: 20-weeks
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Swimming | Control
Number analyzed (Participants) | 52 | 48
millimeters of mercury (mmHg) | 135 (1) | 145 (1)

3. Secondary Outcome: Pressure Wave Reflection
Description: via Augmentation Index
Time Frame: 20-weeks
Measure: Mean (Standard Deviation); unit: % of wave reflection
Arm/Group | Swimming | Control
Number analyzed (Participants) | 52 | 48
% of wave reflection | 25 (2) | 31 (2)

4. Secondary Outcome: Muscular Strength
Description: via Hand Grip Dynamometer
Time Frame: 20-weeks
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Swimming | Control
Number analyzed (Participants) | 52 | 48
kilograms (kg) | 27 (1) | 24 (1)

5. Secondary Outcome: Cardiorespiratory Endurance (Volume of Maximal Oxygen Consumption)
Description: via Cornell Modified Bruce treadmill volume of oxygen consumption maximum (VO2max) test
Time Frame: 20-weeks
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Swimming | Control
Number analyzed (Participants) | 52 | 48
mL/kg/min | 26 (3) | 23 (4)

6. Secondary Outcome: Diastolic Blood Pressure
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Swimming | Control
Number analyzed (Participants) | 52 | 48
millimeters of mercury (mmHg) | 79 (1) | 91 (1)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Swimming | Control
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/48
Other Adverse Events (participants affected / at risk) | 0/52 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT03546270/Prot_SAP_000.pdf